CLINICAL TRIAL: NCT02459769
Title: Exercise Intervention for Lesbian, Gay, Bisexual, and Transgender (LGBT) Cancer Survivors and Caregivers
Brief Title: Exercise Intervention for LGBT Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Charles Kamen, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 56965
Record Dates: First submitted 2015-05-21; First posted 2015-06-02 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dyadic Exercise Intervention (Active Comparator): Progressive walking and resistance exercise treatment, prescribed to both cancer survivors and their caregivers (daily walking and 3 times/week resistance prescription for 6 weeks). Cancer survivor and caregiver are also asked to discuss ways they can support one another in a) remaining adherent to exercise, and b) dealing with stress, including LGBT-specific minority stress.
  Interventions: Behavioral: Exercise for Cancer Patients
- Individual Exercise Intervention (Other): Progressive walking and resistance exercise treatment, prescribed solely to cancer survivors (daily walking and 3 times/week resistance prescription for 6 weeks). The caregiver is told not to change his/her exercise behavior in any way.
  Interventions: Behavioral: Exercise for Cancer Patients

INTERVENTIONS:
Behavioral: Exercise for Cancer Patients — a standardized, daily, 6 week, home-based, progressive exercise program
  Other Names: EXCAP

SUMMARY:
The purpose of this study is to test preliminary efficacy, as well as acceptability and feasibility, of a dyadic exercise intervention, the current study will randomize LGBT cancer survivors and their non-professional caregivers as dyads to either an individual or a dyadic Exercise for Cancer Patients (EXCAP) intervention. The primary outcome assessed will be psychological distress. Analyses will involve pre-post comparisons of outcomes across the study arms, testing the hypothesis that a 6 week, daily, dyadic exercise intervention will result in greater improvements in psychological distress than an individual intervention.

DETAILED DESCRIPTION:
The proposed randomized controlled trial aims to recruit 70 lesbian, gay, bisexual, and transgender (LGBT) cancer survivors who have completed treatment (surgery, radiation, or chemotherapy) within the past 24 months, so as to have a final, evaluable sample of 60 LGBT survivors after attrition. The proposed RCT will also recruit caregivers (broadly defined) of the above cancer survivors. Each recruited cancer survivor will be asked to name a person who they feel provided care (emotional, informational, tangible, etc.) during their cancer experience, with no further strictures placed on this relationship in terms of type or duration. The caregiver will be approached to participate in the RCT. Thus the sample will consist of 70 LGBT survivors (60 evaluable) and their caregivers (140 individuals total/120 evaluable). Recruitment and primary analyses will specifically target the LGBT cancer survivor.

All data will be gathered from participants 21 years of age or older. Participants are cancer survivors who have completed treatments or caregivers of cancer survivors; both survivors and caregivers are able to read and understand English.

ELIGIBILITY:
Inclusion Criteria:

* (Survivors): To be included in the study, cancer survivors must:
* Have had a diagnosis of cancer (any cancer type excluding squamous and basal cell [skin cancers]) and have completed primary surgery, chemotherapy, and/or radiation (those on continued adjuvant treatment are still eligible),
* Identify as lesbian, gay, bisexual, or transgender, or have a same-sex romantic partner,
* Have a caregiver willing to participate in the study (defined as anyone who provided emotional support or tangible assistance during the survivors' cancer experience),
* Be able to read English,
* Be 21 years of age or older, and
* Give written informed consent.
* (Caregivers): Caregivers must:
* Be nominated by a cancer survivor,
* Be able to read English,
* Be 21 years of age or older,
* Give written informed consent.

Exclusion Criteria:

* Have physical limitations (e.g., cardiorespiratory, orthopedic) contraindicating participating in a low- to moderate-intensity home-based walking and progressive resistance program and physical function testing, as assessed by their medical oncologist, their primary care physician, and/or the study medical monitor (or any of these three physicians' designees),
* For caregivers, be currently undergoing active treatment for cancer.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kamen, PhD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dyadic Exercise Intervention for LGBT Survivors; Dyadic Exercise Intervention for Caregivers: Progressive walking and resistance exercise treatment, prescribed to both cancer survivors and their caregivers (daily walking and 3 times/week resistance prescription for 6 weeks). Cancer survivors and caregivers are also asked to discuss ways they can support one another in a) remaining adherent to exercise, and b) dealing with stress, including LGBT-specific minority stress.
  Exercise for Cancer Patients: a standardized, daily, 6 week, home-based, progressive exercise program
- Individual Exercise Intervention for LGBT Cancer Survivors: Progressive walking and resistance exercise treatment, prescribed solely to cancer survivors (daily walking and 3 times/week resistance prescription for 6 weeks). The caregiver is told not to change his/her exercise behavior in any way.
  Exercise for Cancer Patients: a standardized, daily, 6 week, home-based, progressive exercise program
- Individual Caregivers-No Intervention: A caregiver is defined as any individual whom the cancer survivor nominates as having provided emotional support or tangible assistance without pay during the survivor's cancer experience. No restriction will be placed on caregivers in terms of relationship with the cancer survivor; they can be family members, friends, romantic partners, or community members
Period: Overall Study
Arm/Group | Dyadic Exercise Intervention for LGBT Survivors | Individual Exercise Intervention for LGBT Cancer Survivors | Dyadic Exercise Intervention for Caregivers | Individual Caregivers-No Intervention
Started | 34 | 32 | 34 | 33
Completed | 26 | 28 | 25 | 28
Not Completed | 8 | 4 | 9 | 5
Not completed — Withdrawal by Subject | 7 | 4 | 8 | 5
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The above number reflects participants who completed at least the baseline study visit. The number differs from the previous page total as anyone who consented was counted towards the total enrollment number.
Groups:
- Dyadic Exercise Intervention for LGBT Cancer Survivors; Dyadic Exercise Intervention for Caregivers: Progressive walking and resistance exercise treatment, prescribed to both cancer survivors and their caregivers (daily walking and 3 times/week resistance prescription for 6 weeks). Cancer survivors and caregivers are also asked to discuss ways they can support one another in a) remaining adherent to exercise, and b) dealing with stress, including LGBT-specific minority stress.
  Exercise for Cancer Patients: a standardized, daily, 6 week, home-based, progressive exercise program
- Total: Total of all reporting groups
Arm/Group | Dyadic Exercise Intervention for LGBT Cancer Survivors | Individual Exercise Intervention for LGBT Cancer Survivors | Dyadic Exercise Intervention for Caregivers | Individual Caregivers-No Intervention | Total
Number analyzed (Participants) | 32 | 31 | 32 | 31 | 126
Age, Continuous [Mean (Full Range); unit: years] | 56.3 [33 to 78] | 55.5 [28 to 76] | 56.7 [25 to 71] | 54.5 [23 to 77] | 55.7 [23 to 78]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 8 | 13 | 9 | 11 | 41
  Female | 23 | 18 | 23 | 19 | 83
  Transgender Female | 1 | 0 | 0 | 0 | 1
  Transgender Male | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 30 | 31 | 32 | 30 | 123
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 0 | 4
  White | 30 | 31 | 30 | 31 | 122
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 31 | 32 | 31 | 126
Sexual Orientation [Count of Participants; unit: Participants]
  Lesbian or Gay | 30 | 31 | 30 | 26 | 117
  Heterosexual or Straight | 0 | 0 | 1 | 5 | 6
  Bisexual | 1 | 0 | 0 | 0 | 1
  Other | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Psychological Distress
Description: Self-reported psychological distress was measured with the Profile of Mood States (POMS) total score among LGBT cancer survivors. The POMS consists of 30 adjectives that subjects rate on a five-point scale with "1" = "Not at all" and "5" = "Extremely" to describe their moods over the past week. The total score can be calculated by adding the raw scores from tension, depression, anger, fatigue and confusion-focused items and then subtracting the vigour-focused items. This will give a value between -24 and 177, with higher scores indicating higher psychological distress.
Time Frame: Assessed at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Dyadic Exercise Intervention for LGBT Cancer Survivors: Progressive walking and resistance exercise treatment, prescribed to both cancer survivors and their caregivers (daily walking and 3 times/week resistance prescription for 6 weeks). Cancer survivor and caregiver are also asked to discuss ways they can support one another in a) remaining adherent to exercise, and b) dealing with stress, including LGBT-specific minority stress.
  Exercise for Cancer Patients: a standardized, daily, 6 week, home-based, progressive exercise program
Arm/Group | Dyadic Exercise Intervention for LGBT Cancer Survivors | Individual Exercise Intervention for LGBT Cancer Survivors
Number analyzed (Participants) | 32 | 31
score on a scale | 8.89 (22.04) | 6.96 (17.78)

2. Secondary Outcome: Biological Endpoints: Cortisol
Description: The secondary aim is to determine the preliminary effect of EXCAP-PA versus survivor-only EXCAP©® on biological endpoints associated with distress: serum cortisol among LGBT cancer survivors.
Time Frame: Assessed at 8 weeks
Population: Note that only 30 LGBT survivors from the Dyadic Exercise Intervention and only 27 from the Individual Exercise intervention had analyzable blood, which is why the total number of participants differs from other outcome measures.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Dyadic Exercise Intervention for LGBT Cancer Survivors | Individual Exercise Intervention for LGBT Cancer Survivors
Number analyzed (Participants) | 30 | 27
ng/ml | 42.97 (25.83) | 59.20 (49.21)

3. Secondary Outcome: Biological Endpoints: Serum Amyloid A
Description: The secondary aim is to determine the preliminary effect of EXCAP-PA versus survivor-only EXCAP©® on biological endpoints associated with distress: markers of early inflammation serum amyloid A (SAA) among LGBT cancer survivors.
Time Frame: Assessed at 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Dyadic Exercise Intervention for LGBT Cancer Survivors | Individual Exercise Intervention for LGBT Cancer Survivors
Number analyzed (Participants) | 30 | 27
ng/ml | 666.27 (219.98) | 968.26 (1592.59)

4. Secondary Outcome: Biological Endpoints: C-reactive Protein
Description: The secondary aim is to determine the preliminary effect of EXCAP-PA versus survivor-only EXCAP©® on biological endpoints associated with distress: markers of C-reactive protein (CRP) among LGBT cancer survivors.
Time Frame: Assessed at 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Dyadic Exercise Intervention for LGBT Cancer Survivors | Individual Exercise Intervention for LGBT Cancer Survivors
Number analyzed (Participants) | 30 | 27
pg/ml | 860440.91 (2270252.50) | 133590.00 (198748.60)

5. Secondary Outcome: Mechanistic Outcomes: Support
Description: Social support from the care partner was measured with the Dyadic Support Questionnaire (DSQ) among LGBT cancer survivors. The DSQ is an 18-item survey based on four functions of social support (emotional, appraisal, instrumental, and informational support). Nine items measure received social support, that is, support provided by the partner. Items are anchored using a Likert scale ranging from 1 to 5 (from not at all to a great deal). Items were summed to create a scale for received support ranging from 9-45, with higher scores indicating more support.
Time Frame: Assessed at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dyadic Exercise Intervention for LGBT Cancer Survivors | Individual Exercise Intervention for LGBT Cancer Survivors
Number analyzed (Participants) | 32 | 31
score on a scale | 39.46 (7.95) | 39.04 (4.08)

6. Secondary Outcome: Mechanistic Outcomes: Adherence
Description: We also aim to determine the preliminary effect of EXCAP-PA versus survivor-only EXCAP©® on social support from the care partners intervention adherence (actigraphy) among LGBT cancer survivors. The actigraph features a variable epoch length which can be set between 1 to 240 seconds. Software supplied by the manufacturer was used to determine number of minutes of moderate or higher activity during each assessment period.
Time Frame: Assessed at 8 weeks
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Dyadic Exercise Intervention for LGBT Cancer Survivors | Individual Exercise Intervention for LGBT Cancer Survivors
Number analyzed (Participants) | 32 | 31
minutes per day | 12.57 (7.55) | 15.55 (9.60)

7. Other Pre Specified Outcome: Self-Reported Distress Among Caregivers
Description: Self-reported psychological distress among caregivers of LGBT cancer survivors was determined using the Profile of Mood States (POMS) total score. The POMS consists of 30 adjectives that subjects rate on a five-point scale with "1" = "Not at all" and "5" = "Extremely" to describe their moods over the past week. The total score can be calculated by adding the raw scores from tension, depression, anger, fatigue and confusion-focused items and then subtracting the vigour-focused items. This will give a value between -24 and 177, with higher scores indicating higher psychological distress.
Time Frame: Assessed at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Dyadic Exercise Intervention for Caregivers: Progressive walking and resistance exercise treatment, prescribed to both cancer survivors and their caregivers (daily walking and 3 times/week resistance prescription for 6 weeks). Cancer survivor and caregiver are also asked to discuss ways they can support one another in a) remaining adherent to exercise, and b) dealing with stress, including LGBT-specific minority stress.
  Exercise for Cancer Patients: a standardized, daily, 6 week, home-based, progressive exercise program
- Individual Caregivers-No Intervention: Progressive walking and resistance exercise treatment, prescribed solely to cancer survivors (daily walking and 3 times/week resistance prescription for 6 weeks). The caregiver is told not to change his/her exercise behavior in any way.
  Exercise for Cancer Patients: a standardized, daily, 6 week, home-based, progressive exercise program
Arm/Group | Dyadic Exercise Intervention for Caregivers | Individual Caregivers-No Intervention
Number analyzed (Participants) | 32 | 31
score on a scale | 2.65 (16.03) | 6.21 (17.58)

8. Other Pre Specified Outcome: Biological Endpoints of Distress Among Caregivers
Description: An exploratory aim is to determine the preliminary effect of EXCAP-PA versus survivor-only EXCAP©® on biological endpoints associated with distress among caregivers of LGBT cancer survivors: serum cortisol.
Time Frame: Assessed at 8 weeks
Population: Note that only 30 caregivers from the Dyadic Exercise Intervention and only 27 from the Individual Exercise intervention had analyzable blood, which is why the total number of participants differs from other outcome measures.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Dyadic Exercise Intervention for Caregivers | Individual Caregivers-No Intervention
Number analyzed (Participants) | 30 | 27
ng/ml | 68.80 (60.46) | 60.74 (72.42)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Dyadic Exercise Intervention for LGBT Cancer Survivors | Individual Exercise Intervention for LGBT Cancer Survivors | Dyadic Exercise Intervention for Caregivers | Individual Caregivers-No Intervention
All-Cause Mortality (participants affected / at risk) | 3/32 | 2/31 | 1/32 | 1/31
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/31 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/32 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dyadic Exercise Intervention for LGBT Cancer Survivors (N=32) | Individual Exercise Intervention for LGBT Cancer Survivors (N=31) | Dyadic Exercise Intervention for Caregivers (N=32) | Individual Caregivers-No Intervention (N=31)
Serious Adverse Event (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT02459769/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT02459769/ICF_001.pdf